CLINICAL TRIAL: NCT02744573
Title: Evaluation Of The Analgesia Nociception Index vs. Surgical Pleth Index Under General And Regional Anaesthesia And The Effect Of Posture. A Prospective Randomized Controlled Trial.
Brief Title: Evaluation Of The Analgesia Nociception Index vs. Surgical Pleth Index Under General And Regional Anaesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Timo Iden, Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: ANI_SPI
Record Dates: First submitted 2015-12-14; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Pain; Stress; Monitoring
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- General Anaesthesia: ANI and SPI values under general anaesthesia
- Spinal Anaesthesia: ANI and SPI values under spinal anaesthesia
- Spinal Anaesthesia + Sedation: ANI and SPI values under spinal anesthesia in combination with sedation
- Control: ANI and SPI values under no anaesthesia

SUMMARY:
There is a lack of sufficient analgesia monitoring apart from surrogate parameters. The analgesia nociception index (ANI) shall be evaluated under general and regional anaesthesia.

DETAILED DESCRIPTION:
While sophisticated haemodynamic monitoring as well as depth of neuromuscular block and sedation are established in daily clinical routine monitoring of analgesia remains poorly represented. The surgical pleth index (SPI) algorithm takes into account both central and peripheral sympathetic tone via the normalised heart beat interval and the plethysmographic pulse wave amplitude and has been described before. A more detailed investigation on the SPI and its behaviour under a posture maneuver shows the limitation of the device.

Another device developed calculates the "analgesia nociception index" (ANI) by heart rate variability and was launched into the market in 2010. However, the effect of posture - to our knowledge - has not yet been studied. The change of body positioning during surgery is regularly necessary in order to improve surgical access to anatomic structures. These alterations in positioning are known to be accompanied by changes in haemodynamic parameters.

The aim of this study was to evaluate the ANI in patients undergoing elective surgery in lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Body mass index (BMI) < 35 kg m2
* American Society of Anesthesiologists (ASA) status I-III
* Elective urology and gynaecology surgery in lithotomy position
* 15 healthy volunteers were included in the study as a control group

Exclusion Criteria:

* Age < 18 years
* ASA status IV or higher
* BMI ≥ 35 kg m2
* Chronic heart rhythm disorders
* Implanted pacemakers
* Patients with a history of chronic pain and emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of 45 patients ≥ 18 years with a body mass index (BMI) < 35 kg m-2 and an American Society of Anesthesiologists (ASA) status I-III scheduled for elective urology and gynaecology surgery in lithotomy position were randomized. Additionally, 15 volunteers served as a control group under no anaesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ANI vs. SPI | Data will be assessed and collected immediately after completion of each case of surgery.
  Evaluation of the ANI and comparison to SPI (same unit of measure, both ranging between 0-100, no dimension) in patients undergoing elective surgery in lithotomy position. Evaluation and change of ANI and SPI values at pre-defined timepoints: 1) Baseline, 2) before induction of anaesthesia, during 3) intubation or spinal punction, 4) posture maneuver, 5) skin incision 6) surgical suture, 7) post anesthetic care unit stay (arrival).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Grünewald, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Ilies C, Ludwigs J, Gruenewald M, Thee C, Hanf J, Hanss R, Steinfath M, Bein B. The effect of posture and anaesthetic technique on the surgical pleth index. Anaesthesia. 2012 May;67(5):508-513. doi: 10.1111/j.1365-2044.2011.07051.x. Epub 2012 Feb 11. PMID 22324319
- [Background] Boselli E, Daniela-Ionescu M, Begou G, Bouvet L, Dabouz R, Magnin C, Allaouchiche B. Prospective observational study of the non-invasive assessment of immediate postoperative pain using the analgesia/nociception index (ANI). Br J Anaesth. 2013 Sep;111(3):453-9. doi: 10.1093/bja/aet110. Epub 2013 Apr 16. PMID 23592690